CLINICAL TRIAL: NCT03427970
Title: Efficacy of Three-dimensionally Integrated Exercise for Scoliosis in Patients With Adolescent Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing Du, Ph.D, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-18-004
Record Dates: First submitted 2018-01-28; First posted 2018-02-09 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Scoliosis,Idiopathic,Adolescent
MeSH Terms: conditions — Scoliosis | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Control subjects will receive observation for 6 months.
  Interventions: Behavioral: observation
- experimental group (Experimental): Experimental group will perform three-dimensionally integrated exercise for scoliosis for a 60-min period for 1-2 times a week under the guidance of physical therapist in an outpatient clinic, and a 20-min period per day under the supervision of the parents at home.The treatment regimens lasted for 6 months.
  Interventions: Behavioral: three-dimensionally integrated exercise for scoliosis

INTERVENTIONS:
Behavioral: observation — Control group will receive the standard of care according to the Scoliosis Research Society criteria: observation for patients with curves between 10°- 25°.
  Arms: control group
Behavioral: three-dimensionally integrated exercise for scoliosis — Experimental group will receive a modified physiotherapeutic scoliosis specific exercises --the three-dimensionally integrated exercise for scoliosis program, which include auto-correction in 3D, postural correction, breathing training, resistance training, muscle fascia releasing, functional activities, balance training, core stability training, proprioceptive input exercises and patient education. Auto-correction exercise in 3D will combine with specific breathing mode, isometric training to correct abnormal spinal physiological curvatures in sagittal plane, and accompany with wedge pad to modify humpback, waist asymmetry, pelvic rotation in horizontal. While in coronal plane, longitudinal axial stretching, pelvic adjustments will be conducted to reduce the lateral curvature.
  Arms: experimental group

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is one of the most prevalent spinal deformity that may progress sharply during growth. It is recommended that the physiotherapeutic scoliosis-specific exercises should be the first step to treat idiopathic scoliosis to prevent/limit progression of the deformity. Three-dimensionally integrated exercise for scoliosis is based the theory of physiotherapeutic scoliosis specific exercises, and consists of patient education, 3-dimension self-correction, stabilization of the corrected posture and training activity of daily living, combined with neuro-motor control, proprioceptive training, balance training, etc., forming the individual exercise approach for each patient. Nevertheless, the evidence concerning three-dimensionally integrated exercise for scoliosis is inadequate. Therefore, the objective of this study is to determine the effect of three-dimensionally integrated exercise intervention on the change of Cobb angle, angle of trunk rotation(ATR), sagittal profile, and quality of life, compared to standard care for patients with mild AIS.

Informed consent will be obtained from each patient and one of their parents prior to inclusion. Eligible subjects will be randomized by a 1:1 allocation ratio by computer either to the experimental group, in which they will perform three-dimensionally integrated exercise for scoliosis, or the control group, in which they will receive the standard of care with observation according to the Scoliosis Research Society criteria.Blinded assessments at baseline and immediately post 6-month intervention will include radiographic measurement, trunk rotation, sagittal profile and health related quality-of-life.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is one of the most prevalent spinal deformity that may progress sharply during growth. According to the severity of the curve, the major treatment approaches for patient with AIS include exercises, bracing and surgery, to correct, prevent or stop the progression of the deformity.In North America, Scoliosis Research Society (SRS) has been published the standard of care for AIS: patients with curves between 10 and 25° should be observation who are still growing. While in the Europe, the International Scientific Society on Scoliosis Orthopaedic and Rehabilitation Treatment (SOSORT) has recommended that the physiotherapeutic scoliosis-specific exercises should be the first step to treat idiopathic scoliosis to prevent/limit progression of the deformity. Three-dimensionally integrated exercise for scoliosis is based the theory of physiotherapeutic scoliosis specific exercises, and consists of patient education, 3-dimension self-correction, stabilization of the corrected posture and training activity of daily living, combined with neuro-motor control, proprioceptive training, balance training, etc., forming the individual exercise approach for each patient. Nevertheless, the evidence concerning three-dimensionally integrated exercise for scoliosis is inadequate. Therefore, the objective of this study is to determine the effect of three-dimensionally integrated exercise intervention on the change of Cobb angle, angle of trunk rotation(ATR), sagittal profile, and quality of life, compared to standard care for patients with mild AIS.

The present study is a single-center prospective randomised controlled trial conducted at the department of rehabilitation medicine, Xinhua Hospital affiliated to Shanghai Jiao Tong University School of Medicine. The demographic data (height, weight), menarche status for the girls, family history, will be recorded by the physician.

Informed consent will be obtained from each patient and one of their parents prior to inclusion. Eligible subjects will be randomized by a 1:1 allocation ratio by computer either to the experimental group, in which they will perform three-dimensionally integrated exercise for scoliosis, or the control group, in which they will receive the standard of care with observation according to the Scoliosis Research Society criteria. Blinded assessments at baseline and immediately post 6-month intervention will include radiographic measurement, trunk rotation, sagittal profile and health related quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of adolescent idiopathic scoliosis;
* Age from 10 to 16 years;
* A Cobb angle of 10 to 20 degree;
* A Risser sign of 0-3;
* No other treatment which might affect scoliosis.

Exclusion Criteria:

* Non-idiopathic scoliosis, which caused by neuromuscular disorder, vertebral malformation, trauma, tumor, or other diseases;
* Accompanying mental problems, neurological-muscular or rheumatic diseases;
* Previous operation history of spine or lower extremities;
* Previous exercises or brace treatment history;
* Having contraindications to exercise.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Cobb angle | up to 6 months
  It is recommended that curve magnitude of scoliosis is measured using the Cobb method. The Cobb angle will be measured on the standing frontal radiograph according to the Cobb method by the physician specializing in the treatment of scoliosis.

SECONDARY OUTCOMES:
Angle of trunk rotation | up to 6 months
  The angle of trunk rotation will be measured with a Scoliometer. Patients will be asked to bend forward, and the physician will measure the angle of trunk rotation using the Scoliometer.
Sagittal index | up to 6 months
  The Sagittal index (SI) is the sum of plumbline distances from C7 and L3. When SI<60mm,it is considered to be flat black; 60-90mm is in the normal range; >90 mm is considered to kyphosis.
SRS-22 dimensions scores | up to 6 months
  SRS-22 questionnaire is designed for patients with scoliosis specially , which consists of 22 items with 5 dimensions: function/activity, pain, self-Image, mental health, and satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Du, Ph.D, Principal Investigator — Xin Hua Hospital,Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xin Hua Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liang J, Zhou X, Chen N, Li X, Yu H, Yang Y, Song Y, Du Q. Efficacy of three-dimensionally integrated exercise for scoliosis in patients with adolescent idiopathic scoliosis: study protocol for a randomized controlled trial. Trials. 2018 Sep 10;19(1):485. doi: 10.1186/s13063-018-2834-x. PMID 30201050